CLINICAL TRIAL: NCT04851899
Title: Efficacy of a Microalgae Extract PhaeoSOL Combined With Natural Stimulant on Cognitive Function and Gaming Performance of Video Gamers
Acronym: PHAEOSOL-TWO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microphyt (Industry)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB2021-0219
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Cognitive Function; Video Gamers
Keywords: Fucoxanthin; Microalgae; Gaming performance; E-sports; Cognitive performance; Energy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose Phaeosol group (Experimental): 1 Phaeosol softgel of 440mg/day and 1 placebo softgel of 440mg/day look like softgel of Phaeosol product) + 1 capsule of 440mg/day of natural stimulant
  Interventions: Dietary Supplement: Phaeosol low dose
- High dose Phaeosol group (Experimental): 2 Phaeosol softgels of 440mg/day + 1 capsule of 440mg/day of natural stimulant
  Interventions: Dietary Supplement: Phaeosol high dose
- Placebo group (Placebo Comparator): 2 placebo softgels of 440mg/day (look like softgel of Phaeosol product) + 1 capsule of 440mg/day containing Microcellulose (look like capsule of natural stimulant)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phaeosol low dose — 1 Phaeosol softgel of 440mg/day and 1 placebo softgel of 500mg/day (look like softgel of Phaeosol product) + 1 capsule of 440mg/day of natural stimulant Subjects were instructed to take the study supplement or placebo once daily for 1 months (±2 days). The first and the last doses will be administered at the clinical site during Visit 2 (Experiment 1) and Visit 3 (Experiment 2, respectively).
  Arms: Low dose Phaeosol group
Dietary Supplement: Phaeosol high dose — 2 Phaeosol softgels of 440mg/day + 1 capsule of 440mg/day of natural stimulant. Subjects were instructed to take the study supplement or placebo once daily for 1 months (±2 days). The first and the last doses will be administered at the clinical site during Visit 2 (Experiment 1) and Visit 3 (Experiment 2, respectively).
  Arms: High dose Phaeosol group
Dietary Supplement: Placebo — 2 placebo softgels of 440mg/day (look like softgel of Phaeosol product) + 1 capsule of 500mg/day containing Microcellulose (look like capsule of natural stimulant). Subjects were instructed to take the study supplement or placebo once daily for 1 months (±2 days). The first and the last doses will be administered at the clinical site during Visit 2 (Experiment 1) and Visit 3 (Experiment 2, respectively).
  Arms: Placebo group

SUMMARY:
Considering the important growing development of gaming in the world, this research area has developed considerably over the last few years. Even if it seems to be well admitted that video gamers showed better cognitive functions (e.g. visual selective attention, cognitive flexibility, task switching) parameters compared to non video gamers there is a constant concern for optimizing performance as for all other kind of athletes. However to our knowledge, only one randomized controlled trial have investigated the potential benefits of dietary supplementation on cognitive function and performance in video gamers. The use of microalgea as molecule of interest sources is a recent promising approach also to meet societal challenge as the maintain of biodiversity/landscape.

Thus, the purpose of this study is to examine whether acute (single-dose) and chronic (1 month) supplementation of Microphyt's phaeosol ingredients (BrainPhyt) ingested with or without a natural stimulant, would affect cognitive function and gaming performance in experienced video gamers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women;
2. Between 18 and 40 years;
3. Self-reported history of playing video games for 5 or more hours per week for 6 months prior to screening;
4. BMI between 18 and 34.9 Kg/m2 ;
5. Subjects agreed to supply their own operator-oriented action or strategy video game that they had played at least 21 times over the last 3 months;
6. No recent ingestion (<2weeks) of dietary supplement that affect cognitive function;
7. Be able to give written informed consent and to consume the investigational product daily for the duration of the study;
8. Is free-living (living in a private home, alone or with family, and able to maintain their health and hygiene without assistance)
9. Willing to maintain consistent sleep duration the evening before study visits.
10. Are agreed to continue their patterned use of the game between study visits

Exclusion Criteria:

1. refrain from caffeine and alcohol for 12 hours prior to each study visits;
2. consume dietary supplements that may affect cognition and/or with a stimulant effect (e.g. guarana, cocoa, ginseng, bacopa, Gingko biloba, guayusa, yerba mate, energy drinks, other products containing fucoxanthin) at least 7 days before Visit 2 ;
3. are women who are pregnant, breastfeeding, or wish to become pregnant during the study;
4. have an untreated psychotic or major depressive disorder or any history of cognitive deficit;
5. have an uncontrolled hypertension/diabetes/thyroid/heart disease disease, cancer etc.);
6. have a significant neurological disease;
7. have planned major changes in lifestyle (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
8. have a history within previous 12 months of alcohol or substance abuse;
9. have known allergy to any of the ingredients in the supplement product
10. are not willing to supply their own gaming system and/or game

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Reaction time | From week 0 to week 4
  Change in reaction time - Light tracking test
General attention | From week 0 to week 4
  Change in general attention score - Go no go task test
Sustained attention | From week 0 to week 4
  Change in sustained attention score - Psychomotor vigilance task test
Attention shifting | From week 0 to week 4
  Change in attention shifting score - Berg-Washington card sorting task test

SECONDARY OUTCOMES:
Gaming performance | From week 0 to week 4
  Change in gaming performance score from 0 to 100 - Higher scores mean a better outcome
Mood state | From week 0 to week 4
  Change in Mood state questionnaire score from 0 to 100 - Higher scores mean a better outcome - Profil of Mood state questionnaire
Sleep quality | From week 0 to week 4
  Change in sleep quality questionnaire score from 0 to 100 - Higher scores mean a better outcome
Eyes irritability | From week 0 to week 4
  Change in eyes irritability score -Visual analogic scale from 0 to 100 - Higher scores mean a worse outcome
Global fatigue | From week 0 to week 4
  Change in global fatigue score - Visual analogic scale from 0 to 100 - higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kreider, Professor, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leonard M, Maury J, Dickerson B, Gonzalez DE, Kendra J, Jenkins V, Nottingham K, Yoo C, Xing D, Ko J, Pradelles R, Faries M, Kephart W, Sowinski R, Rasmussen CJ, Kreider RB. Effects of Dietary Supplementation of a Microalgae Extract Containing Fucoxanthin Combined with Guarana on Cognitive Function and Gaming Performance. Nutrients. 2023 Apr 15;15(8):1918. doi: 10.3390/nu15081918. PMID 37111136